CLINICAL TRIAL: NCT05445921
Title: Stellate Ganglion Block for the Treatment of COVID-19-Induced Olfactory Dysfunction: A Prospective Pilot Study
Brief Title: Stellate Ganglion Block for COVID-19-Induced Olfactory Dysfunction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Nyssa Farrell, Nyssa Farrell, MD, Assistant Professor, Department of Otolaryngology - Head and Neck Surgery, Division of Rhinology and Anterior Skull Base Surgery, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202207170
Record Dates: First submitted 2022-07-02; First posted 2022-07-06 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2023-10

CONDITIONS: Anosmia; Hyposmia; Parosmia; Olfactory Disorder
Keywords: COVID-19
MeSH Terms: conditions — Anosmia; Olfaction Disorders; COVID-19 | interventions — Mepivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Stellate Ganglion Block (Experimental): The ultrasound guided stellate ganglion blocks will be performed by a pain management specialist with extensive experience performing these blocks. The first SGB at the initial visit will be performed on the right side, and the second SGB will be on the left side 5-10 days after the first SGB, given that the patient tolerated the first SGB.
  Interventions: Drug: Stellate Ganglion Block

INTERVENTIONS:
Drug: Stellate Ganglion Block — The stellate ganglion will be identified using ultrasound guidance, and after a test does of 1% lidocaine, 1% mepivacaine will be injected near the stellate ganglion.
  Other Names: mepivacaine

SUMMARY:
Chronic olfactory dysfunction from the COVID-19 pandemic is a growing public health crisis with up to 1.2 million people in the Unites States affected. Olfactory dysfunction impacts one's quality of life significantly by decreasing the enjoyment of foods, creating environmental safety concerns, and affecting one's ability to perform certain jobs. Olfactory dysfunction is also an independent predictor of anxiety, depression, and even mortality. While the pandemic has increased the interest by the scientific community in combating the burgeoning health crisis, few effective treatments currently exist for olfactory dysfunction. Furthermore, patients impacted by "long COVID," or chronic symptoms after an acute COVID-19 infection, experience impairments other than olfactory and gustatory dysfunction, such as chronic dyspnea, impaired memory and concentration, and severe fatigue. These symptoms have been hypothesized to be a result of sympathetic positive feedback loops and dysautonomia. Stellate ganglion blocks have been proposed to treat this hyper-sympathetic activation by blocking the sympathetic neuronal firing and resetting the balance of the autonomic nervous system. Studies prior to the COVID-19 pandemic have supported a beneficial effect of stellate ganglion blocks on olfactory dysfunction, and recent news reports and a published case series have described a dramatic benefit in both olfactory function and other long COVID symptoms in patients receiving stellate ganglion blocks. Therefore, we propose a single cohort prospective study to generate pilot data on the efficacy and safety of sequential stellate ganglion blocks for the treatment of COVID-19-induced olfactory dysfunction and other long COVID symptoms.

DETAILED DESCRIPTION:
One of the hallmark symptoms of infection with SARS-CoV-2 is olfactory dysfunction, and it is estimated that up to 1.2 million people in the United States will experience chronic olfactory dysfunction from the COVID-19 pandemic. While the majority of patients recover from COVID dysosmia, up to 15%-25% have long-term hyposmia. Olfactory impairment can take the form of hyposmia (diminished sense of smell), anosmia (absent sense of smell), or parosmia (distorted sense of smell). Etiologies of olfactory dysfunction include post-viral, traumatic, inflammatory (e.g., chronic rhinosinusitis), neurodegenerative (e.g., Parkinson's disease), and congenital, among others. Prior to the pandemic, post-viral anosmia was the most common cause of olfactory dysfunction, which has further increased as the dominant etiology as a result of COVID-19. The proposed pathophysiologic mechanisms of chronic COVID-19-induced olfactory dysfunction include inflammatory cytokine release, damage to the supporting environment of the olfactory epithelium, and retrograde propagation to higher order neurons. A unique feature of COVID-19-associated olfactory dysfunction is the high rate of persistent parosmia. In one study of 222 patients with COVID-19-associated olfactory dysfunction, 148 (67%) of these patients experienced parosmia at some point. Of the 148 patients with parosmia at any point, 84 (57%) had persistent parosmia after a mean of 6.5 months, distinguishing COVID-19-induced olfactory dysfunction from any other etiologies of olfactory dysfunction. Patients with olfactory dysfunction have decreased quality-of-life and describe their life as if "living in a box." These patients have concern for environmental safety, decreased enjoyment of their food, depression, anxiety, and even higher risk of mortality. The COVID-19 pandemic has highlighted the importance of the sense of olfaction, however, there is a scarcity of effective treatments for olfactory dysfunction. Furthermore, chronic olfactory dysfunction is just one of the constellation of symptoms included in "long COVID," or persistent symptoms after recovery from acute illness due to COVID-19. Other symptoms of long COVID include fatigue, dyspnea, cough, and impaired memory and concentration, among many others.These chronic symptoms are hypothesized to be, at least in part, a result of sympathetic hyperactivity resulting in positive feedback loops. Therefore, the stellate ganglion block, which inhibits the sympathetic nervous system, is hypothesized to reset the balance of the autonomic nervous system and provide relief for long COVID symptoms, including olfactory dysfunction.

Treatment No standard of care treatment for post-viral olfactory dysfunction exists. The most commonly used treatment for post-viral olfactory dysfunction is olfactory training; however, a large proportion of patients do not receive benefit and continue to have persistent symptoms. A multitude of other therapies have been tried with minimal success, including theophylline, vitamin A, sodium citrate, and intranasal insulin. As a result, there is a critical need for the development of a novel intervention to address the large volume of patients with olfactory dysfunction as a result of the COVID-19 pandemic.

The stellate ganglion block (SGB) involves an ultrasound-guided injection of a local anesthetic to inhibit the stellate ganglion. The SGB is proposed to inhibit the sympathetic neural connections within the head, neck, and upper extremity, improve regional blood flow, reduce adrenal hormone concentration, and even reestablish circadian rhythms through modulation of melatonin. The SGB has been used successfully in a multitude of disorders, including post-traumatic stress disorder, cluster headache, complex regional pain syndrome, and peripheral vascular disease.

The SGB was first proposed to treat olfactory dysfunction by Lee et al in 2003, where 38 post-viral olfactory dysfunction participants were treated with SGB and 13 participants remained untreated as controls. Subjective olfactory function improved in 27 (71%) of the treated participants compared to zero (0%) of the controls. Olfactory perception was improved significantly in the SGB group assessed both by the butanol threshold test and odor identification test. There were no complications of SGB in the 38 treated participants. Another study in 2007 by Moon et al found that in 13 participants with various etiologies of olfactory dysfunction, seven (54%) demonstrated improvement with repeated SGBs. The same group conducted a study published in 2013 looking at the long-term results of SGB in treating olfactory dysfunction from various etiologies. Of 37 participants with olfactory dysfunction unresponsive to oral or intranasal steroids who underwent SGB, 15 (41%) were determined to be responsive and 22 (59%) unresponsive to the treatment. Importantly, the responsive group had a mean duration of olfactory dysfunction of 1.6 years vs. a mean duration of olfactory dysfunction of 4 years in the unresponsive group. The study found that in those who respond to SGB, the beneficial effects on olfaction last at least 5 years. Of the 37 treated participants there was only 1 who experienced a complication, which was a temporary brachial plexus block.

Most recently, anecdotal news reports and a published case series point to a possible beneficial effect of SGB on both chronic COVID-19-induced olfactory dysfunction and various other long COVID symptoms. A published case series by Liu et al describes two patients who underwent SGB for long COVID symptoms, including olfactory dysfunction. SGB was performed on the right side then either one or two days later to the left side. Both patients reported significant and durable improvement in symptoms, including fatigue, "brain fog," and olfactory and gustatory dysfunction that persisted at 60-day follow-up. Nearly all other long COVID symptoms, including cough, chest pain, heart palpitations, and orthostatic dizziness, also improved at the one week and two-month follow-up time points. The authors concluded that although the sample size is limited, SGB may have a significant impact on the dysautonomia caused by COVID-19 and improve long COVID symptoms, giving rationale to conduct a larger study. Therefore, we propose a single cohort prospective study to generate pilot data on the effectiveness and safety of sequential stellate ganglion blocks for the treatment of COVID-19-induced olfactory dysfunction and other long COVID symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 to 70
2. Diagnosis of COVID at least 12 months prior to study enrollment with self-reported olfactory dysfunction
3. Objective olfactory dysfunction due to COVID-19 that has persisted despite viral recovery, as defined by the UPSIT (≤ 34 in women, ≤ 33 in men)
4. Ability to read, write, and understand English

Exclusion Criteria:

1. History of smell loss prior to COVID-19 infection
2. History of conditions known to impact olfactory function:

   1. Chronic rhinosinusitis
   2. History of prior sinonasal or skull base surgery
   3. Neurodegenerative disorders (Parkinson's disease, Huntington's disease, Amyotrophic lateral sclerosis, Lewy body dementia, frontotemporal dementia)
3. Currently using concomitant therapies specifically for the treatment of olfactory dysfunction
4. Inability to tolerate a needle injection into the neck
5. History of coexisting conditions that make SGB contraindicated:

   1. Unilateral vocal cord paralysis
   2. Severe COPD (FEV1 between 30-50% of predicted)
   3. Recent myocardial infarction within the last year
   4. Glaucoma
   5. Cardiac conduction block of any degree
6. Currently taking blood thinners or antiplatelet agents
7. Allergy to local anesthetic
8. Inability to extend the neck for any reason (e.g., severe arthritis)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine/Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khan AM, Kallogjeri D, Piccirillo JF. Growing Public Health Concern of COVID-19 Chronic Olfactory Dysfunction. JAMA Otolaryngol Head Neck Surg. 2022 Jan 1;148(1):81-82. doi: 10.1001/jamaoto.2021.3379. PMID 34792577
- [Background] Hintschich CA, Fischer R, Hummel T, Wenzel JJ, Bohr C, Vielsmeier V. Persisting olfactory dysfunction in post-COVID-19 is associated with gustatory impairment: Results from chemosensitive testing eight months after the acute infection. PLoS One. 2022 Mar 23;17(3):e0265686. doi: 10.1371/journal.pone.0265686. eCollection 2022. PMID 35320821
- [Background] Fortunato F, Martinelli D, Iannelli G, Milazzo M, Farina U, Di Matteo G, De Nittis R, Ascatigno L, Cassano M, Lopalco PL, Prato R. Self-reported olfactory and gustatory dysfunctions in COVID-19 patients: a 1-year follow-up study in Foggia district, Italy. BMC Infect Dis. 2022 Jan 22;22(1):77. doi: 10.1186/s12879-022-07052-8. PMID 35065619
- [Background] Welge-Lussen A, Wolfensberger M. Olfactory disorders following upper respiratory tract infections. Adv Otorhinolaryngol. 2006;63:125-132. doi: 10.1159/000093758. PMID 16733337
- [Background] Seiden AM. Postviral olfactory loss. Otolaryngol Clin North Am. 2004 Dec;37(6):1159-66. doi: 10.1016/j.otc.2004.06.007. PMID 15563908
- [Background] Cazzolla AP, Lovero R, Lo Muzio L, Testa NF, Schirinzi A, Palmieri G, Pozzessere P, Procacci V, Di Comite M, Ciavarella D, Pepe M, De Ruvo C, Crincoli V, Di Serio F, Santacroce L. Taste and Smell Disorders in COVID-19 Patients: Role of Interleukin-6. ACS Chem Neurosci. 2020 Sep 2;11(17):2774-2781. doi: 10.1021/acschemneuro.0c00447. Epub 2020 Aug 19. PMID 32786309
- [Background] Chang K, Kallogjeri D, Piccirillo J, House SL, Turner J, Schneider J, Farrell NF. Nasal inflammatory profile in patients with COVID-19 olfactory dysfunction. Int Forum Allergy Rhinol. 2022 Jul;12(7):952-954. doi: 10.1002/alr.22939. Epub 2022 Jan 10. No abstract available. PMID 34890110
- [Background] Bryche B, St Albin A, Murri S, Lacote S, Pulido C, Ar Gouilh M, Lesellier S, Servat A, Wasniewski M, Picard-Meyer E, Monchatre-Leroy E, Volmer R, Rampin O, Le Goffic R, Marianneau P, Meunier N. Massive transient damage of the olfactory epithelium associated with infection of sustentacular cells by SARS-CoV-2 in golden Syrian hamsters. Brain Behav Immun. 2020 Oct;89:579-586. doi: 10.1016/j.bbi.2020.06.032. Epub 2020 Jul 3. PMID 32629042
- [Background] Han AY, Mukdad L, Long JL, Lopez IA. Anosmia in COVID-19: Mechanisms and Significance. Chem Senses. 2020 Jun 17:bjaa040. doi: 10.1093/chemse/bjaa040. Online ahead of print. PMID 32556089
- [Background] Lerner DK, Garvey KL, Arrighi-Allisan AE, Filimonov A, Filip P, Shah J, Tweel B, Del Signore A, Schaberg M, Colley P, Govindaraj S, Iloreta AM. Clinical Features of Parosmia Associated With COVID-19 Infection. Laryngoscope. 2022 Mar;132(3):633-639. doi: 10.1002/lary.29982. Epub 2021 Dec 13. PMID 34870334
- [Background] Keller A, Malaspina D. Hidden consequences of olfactory dysfunction: a patient report series. BMC Ear Nose Throat Disord. 2013 Jul 23;13(1):8. doi: 10.1186/1472-6815-13-8. PMID 23875929
- [Background] Santos DV, Reiter ER, DiNardo LJ, Costanzo RM. Hazardous events associated with impaired olfactory function. Arch Otolaryngol Head Neck Surg. 2004 Mar;130(3):317-9. doi: 10.1001/archotol.130.3.317. PMID 15023839
- [Background] Pang NY, Song HJJMD, Tan BKJ, Tan JX, Chen ASR, See A, Xu S, Charn TC, Teo NWY. Association of Olfactory Impairment With All-Cause Mortality: A Systematic Review and Meta-analysis. JAMA Otolaryngol Head Neck Surg. 2022 May 1;148(5):436-445. doi: 10.1001/jamaoto.2022.0263. PMID 35389456
- [Background] Aiyegbusi OL, Hughes SE, Turner G, Rivera SC, McMullan C, Chandan JS, Haroon S, Price G, Davies EH, Nirantharakumar K, Sapey E, Calvert MJ; TLC Study Group. Symptoms, complications and management of long COVID: a review. J R Soc Med. 2021 Sep;114(9):428-442. doi: 10.1177/01410768211032850. Epub 2021 Jul 15. PMID 34265229
- [Background] Fischer L, Barop H, Ludin SM, Schaible HG. Regulation of acute reflectory hyperinflammation in viral and other diseases by means of stellate ganglion block. A conceptual view with a focus on Covid-19. Auton Neurosci. 2022 Jan;237:102903. doi: 10.1016/j.autneu.2021.102903. Epub 2021 Nov 10. PMID 34894589
- [Background] Addison AB, Wong B, Ahmed T, Macchi A, Konstantinidis I, Huart C, Frasnelli J, Fjaeldstad AW, Ramakrishnan VR, Rombaux P, Whitcroft KL, Holbrook EH, Poletti SC, Hsieh JW, Landis BN, Boardman J, Welge-Lussen A, Maru D, Hummel T, Philpott CM. Clinical Olfactory Working Group consensus statement on the treatment of postinfectious olfactory dysfunction. J Allergy Clin Immunol. 2021 May;147(5):1704-1719. doi: 10.1016/j.jaci.2020.12.641. Epub 2021 Jan 13. PMID 33453291
- [Background] Kang CK, Oh ST, Chung RK, Lee H, Park CA, Kim YB, Yoo JH, Kim DY, Cho ZH. Effect of stellate ganglion block on the cerebrovascular system: magnetic resonance angiography study. Anesthesiology. 2010 Oct;113(4):936-44. doi: 10.1097/ALN.0b013e3181ec63f5. PMID 20823762
- [Background] Treggiari MM, Romand JA, Martin JB, Reverdin A, Rufenacht DA, de Tribolet N. Cervical sympathetic block to reverse delayed ischemic neurological deficits after aneurysmal subarachnoid hemorrhage. Stroke. 2003 Apr;34(4):961-7. doi: 10.1161/01.STR.0000060893.72098.80. Epub 2003 Mar 20. PMID 12649526
- [Background] Mulvaney SW, McLean B, de Leeuw J. The use of stellate ganglion block in the treatment of panic/anxiety symptoms with combat-related post-traumatic stress disorder; preliminary results of long-term follow-up: a case series. Pain Pract. 2010 Jul-Aug;10(4):359-65. doi: 10.1111/j.1533-2500.2010.00373.x. Epub 2010 Apr 20. PMID 20412504
- [Background] Lipov EG, Joshi JR, Sanders S, Slavin KV. A unifying theory linking the prolonged efficacy of the stellate ganglion block for the treatment of chronic regional pain syndrome (CRPS), hot flashes, and posttraumatic stress disorder (PTSD). Med Hypotheses. 2009 Jun;72(6):657-61. doi: 10.1016/j.mehy.2009.01.009. Epub 2009 Feb 23. PMID 19237252
- [Background] Liu LD, Duricka DL. Stellate ganglion block reduces symptoms of Long COVID: A case series. J Neuroimmunol. 2022 Jan 15;362:577784. doi: 10.1016/j.jneuroim.2021.577784. Epub 2021 Dec 8. PMID 34922127
- [Background] Doty RL, Shaman P, Dann M. Development of the University of Pennsylvania Smell Identification Test: a standardized microencapsulated test of olfactory function. Physiol Behav. 1984 Mar;32(3):489-502. doi: 10.1016/0031-9384(84)90269-5. PMID 6463130
- [Background] Doty RL. Office procedures for quantitative assessment of olfactory function. Am J Rhinol. 2007 Jul-Aug;21(4):460-73. doi: 10.2500/ajr.2007.21.3043. PMID 17882917
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Dunlop BW, Gray J, Rapaport MH. Transdiagnostic Clinical Global Impression Scoring for Routine Clinical Settings. Behav Sci (Basel). 2017 Jun 27;7(3):40. doi: 10.3390/bs7030040. PMID 28653978
- [Background] McLean B. Safety and Patient Acceptability of Stellate Ganglion Blockade as a Treatment Adjunct for Combat-Related Post-Traumatic Stress Disorder: A Quality Assurance Initiative. Cureus. 2015 Sep 10;7(9):e320. doi: 10.7759/cureus.320. PMID 26487996
- See also: The Efficacy of Stellate Ganglion Block in Olfactory Disorder Following Upper Respiratory Tract Infection — https://www.kjorl.org/journal/view.php?number=2604
- See also: The Efficacy of Stellate Ganglion Block in Sensorineural Anosmia Patients Unresponsive to Steroid Therapy — https://www.epain.org/journal/view.html?volume=20&number=2&spage=154

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stellate Ganglion Block
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Stellate Ganglion Block
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression - Improvement (CGI-I) Score
Description: Participants will be asked about their change in olfactory dysfunction on a 7-point Likert scale from much better to much worse.
Time Frame: 5-10 days post SGB #1 and 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Stellate Ganglion Block
Number analyzed (Participants) | 20
Participants
  CGI-I for Smell Loss at 1 Week: About the Same | 12
  CGI-I for Smell Loss at 1 Week: Slightly Better | 8
  CGI-I for Smell Loss at 1 Week: Moderately Better | 0
  CGI-I for Smell Loss at 1 Week: Much Better | 0
  CGI-I for Smell Loss at 1 Month: About the Same | 10
  CGI-I for Smell Loss at 1 Month: Slightly Better | 6
  CGI-I for Smell Loss at 1 Month: Moderately Better | 3
  CGI-I for Smell Loss at 1 Month: Much Better | 1
  CGI-I for Smell Distortion at 1 Week: About the Same | 11
  CGI-I for Smell Distortion at 1 Week: Slightly Better | 9
  CGI-I for Smell Distortion at 1 Week: Moderately Better | 0
  CGI-I for Smell Distortion at 1 Week: Much Better | 0
  CGI-I for Smell Distortion at 1 Month: About the Same | 11
  CGI-I for Smell Distortion at 1 Month: Slightly Better | 6
  CGI-I for Smell Distortion at 1 Month: Moderately Better | 2
  CGI-I for Smell Distortion at 1 Month: Much Better | 1
  CGI-I for Taste Loss at 1 Week: About the Same | 15
  CGI-I for Taste Loss at 1 Week: Slightly Better | 4
  CGI-I for Taste Loss at 1 Week: Moderately Better | 1
  CGI-I for Taste Loss at 1 Week: Much Better | 0
  CGI-I for Taste Loss at 1 Month: About the Same | 14
  CGI-I for Taste Loss at 1 Month: Slightly Better | 3
  CGI-I for Taste Loss at 1 Month: Moderately Better | 2
  CGI-I for Taste Loss at 1 Month: Much Better | 1
  CGI-I for Taste Distortion at 1 Week: About the Same | 13
  CGI-I for Taste Distortion at 1 Week: Slightly Better | 6
  CGI-I for Taste Distortion at 1 Week: Moderately Better | 1
  CGI-I for Taste Distortion at 1 Week: Much Better | 0
  CGI-I for Taste Distortion at 1 Month: About the Same | 12
  CGI-I for Taste Distortion at 1 Month: Slightly Better | 5
  CGI-I for Taste Distortion at 1 Month: Moderately Better | 2
  CGI-I for Taste Distortion at 1 Month: Much Better | 1

2. Secondary Outcome: University of Pennsylvania Smell Identification Test (UPSIT)
Description: Participants will complete the 40-item scratch and sniff UPSIT and mean change will be assessed.
  The UPSIT has a minimum score of 0 and maximum score of 40 with lower scores indicating a greater degree of impairment. An UPSIT score of >33 for men and >34 for women is considered normosmic, and the minimal clinically important difference is a change of 4 points.
Time Frame: baseline, 5-10 days, and 1 month
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Stellate Ganglion Block
Number analyzed (Participants) | 20
units on a scale
  UPSIT at Baseline | 16.5 [4 to 32]
  UPSIT at 1 Week | 21 [10 to 31]
  UPSIT at 1 Month | 22.5 [10 to 35]

3. Secondary Outcome: Olfactory Dysfunction Outcomes Rating (ODOR)
Description: Participants will be asked to complete the ODOR, which is a patient-reported outcome measure assessing physical problems, functional limitations, and emotional consequences of olfactory dysfunction.
  The ODOR has a minimum score of 0 and a maximum score of 112 with higher scores indicating a greater degree of impairment and limitation. The minimal clinically important difference is a change of 15 points.
Time Frame: baseline, 5-10 days post SGB #1, and 1 month
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Stellate Ganglion Block
Number analyzed (Participants) | 20
score on a scale
  ODOR at Baseline | 62 [16 to 85]
  ODOR at 1 Week | 57 [13 to 82]
  ODOR at 1 Month | 50.5 [2 to 75]

4. Secondary Outcome: Clinical Global Impression - Severity (CGI-S) Score
Description: Participants will be asked about the severity of their olfactory dysfunction (and gustatory dysfunction) on a 5-point Likert scale from no smell loss to severe smell loss.
Time Frame: baseline, 5-10 days, and 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Stellate Ganglion Block
Number analyzed (Participants) | 20
Participants
  CGI-S for Smell Loss at Baseline: No Problem | 0
  CGI-S for Smell Loss at Baseline: Very Mild Problem | 1
  CGI-S for Smell Loss at Baseline: Mild Problem | 2
  CGI-S for Smell Loss at Baseline: Moderate Problem | 5
  CGI-S for Smell Loss at Baseline: Severe Problem | 12
  CGI-S for Smell Loss at 1 Week: No Problem | 0
  CGI-S for Smell Loss at 1 Week: Very Mild Problem | 3
  CGI-S for Smell Loss at 1 Week: Mild Problem | 2
  CGI-S for Smell Loss at 1 Week: Moderate Problem | 8
  CGI-S for Smell Loss at 1 Week: Severe Problem | 7
  CGI-S for Smell Loss at 1 Month: No Problem | 0
  CGI-S for Smell Loss at 1 Month: Very Mild Problem | 5
  CGI-S for Smell Loss at 1 Month: Mild Problem | 1
  CGI-S for Smell Loss at 1 Month: Moderate Problem | 9
  CGI-S for Smell Loss at 1 Month: Severe Problem | 5
  CGI-S for Smell Distortion at Baseline: No Problem | 1
  CGI-S for Smell Distortion at Baseline: Very Mild Problem | 1
  CGI-S for Smell Distortion at Baseline: Mild Problem | 1
  CGI-S for Smell Distortion at Baseline: Moderate Problem | 5
  CGI-S for Smell Distortion at Baseline: Severe Problem | 12
  CGI-S for Smell Distortion at 1 Week: No Problem | 1
  CGI-S for Smell Distortion at 1 Week: Very Mild Problem | 1
  CGI-S for Smell Distortion at 1 Week: Mild Problem | 4
  CGI-S for Smell Distortion at 1 Week: Moderate Problem | 4
  CGI-S for Smell Distortion at 1 Week: Severe Problem | 10
  CGI-S for Smell Distortion at 1 Month: No Problem | 3
  CGI-S for Smell Distortion at 1 Month: Very Mild Problem | 1
  CGI-S for Smell Distortion at 1 Month: Mild Problem | 2
  CGI-S for Smell Distortion at 1 Month: Moderate Problem | 5
  CGI-S for Smell Distortion at 1 Month: Severe Problem | 9
  CGI-S for Taste Loss at Baseline: No Problem | 0
  CGI-S for Taste Loss at Baseline: Very Mild Problem | 3
  CGI-S for Taste Loss at Baseline: Mild Problem | 2
  CGI-S for Taste Loss at Baseline: Moderate Problem | 4
  CGI-S for Taste Loss at Baseline: Severe Problem | 11
  CGI-S for Taste Loss at 1 Week: No Problem | 0
  CGI-S for Taste Loss at 1 Week: Very Mild Problem | 4
  CGI-S for Taste Loss at 1 Week: Mild Problem | 2
  CGI-S for Taste Loss at 1 Week: Moderate Problem | 5
  CGI-S for Taste Loss at 1 Week: Severe Problem | 9
  CGI-S for Taste Loss at 1 Month: No Problem | 0
  CGI-S for Taste Loss at 1 Month: Very Mild Problem | 5
  CGI-S for Taste Loss at 1 Month: Mild Problem | 2
  CGI-S for Taste Loss at 1 Month: Moderate Problem | 7
  CGI-S for Taste Loss at 1 Month: Severe Problem | 6
  CGI-S for Taste Distortion at Baseline: No Problem | 2
  CGI-S for Taste Distortion at Baseline: Very Mild Problem | 2
  CGI-S for Taste Distortion at Baseline: Mild Problem | 1
  CGI-S for Taste Distortion at Baseline: Moderate Problem | 3
  CGI-S for Taste Distortion at Baseline: Severe Problem | 12
  CGI-S for Taste Distortion at 1 Week: No Problem | 2
  CGI-S for Taste Distortion at 1 Week: Very Mild Problem | 3
  CGI-S for Taste Distortion at 1 Week: Mild Problem | 1
  CGI-S for Taste Distortion at 1 Week: Moderate Problem | 5
  CGI-S for Taste Distortion at 1 Week: Severe Problem | 9
  CGI-S for Taste Distortion at 1 Month: No Problem | 3
  CGI-S for Taste Distortion at 1 Month: Very Mild Problem | 2
  CGI-S for Taste Distortion at 1 Month: Mild Problem | 2
  CGI-S for Taste Distortion at 1 Month: Moderate Problem | 6
  CGI-S for Taste Distortion at 1 Month: Severe Problem | 7

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: Adverse events were reported per injection. Since all participants received two injections, there were a total of 40 possible reported events for each particular adverse event.
Arm/Group | Stellate Ganglion Block
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stellate Ganglion Block (N=20)
Horner syndrome (Nervous system disorders) | 20
Hoarseness (Nervous system disorders) | 9
Globus (Nervous system disorders) | 7
Brief lightheadedness (Cardiac disorders) | 5
Numbness of the face (Nervous system disorders) | 4
Mild shortness of breath (Respiratory, thoracic and mediastinal disorders) | 4
Nasal congestion (General disorders) | 3
Pain at the injection site (General disorders) | 3
Fatigue (General disorders) | 3
Cough (General disorders) | 1
Weakness of the arm (Nervous system disorders) | 1
Weakness of the neck/back (General disorders) | 1
Tightness of the back (General disorders) | 1
Arm heaviness (General disorders) | 1
Bruising of the injection site (General disorders) | 1
Chest heaviness (General disorders) | 1
Headache (General disorders) | 1
Palpitations (General disorders) | 1
Tightness of the shoulder (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT05445921/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT05445921/ICF_001.pdf